CLINICAL TRIAL: NCT04927637
Title: A Pilot Study to Evaluate Single Dose Indocyanine Green 24 Hours Prior to Operative Treatment of Orthopaedic Infection
Brief Title: ICG 24h Prior to Operative Treatment of Orthopaedic Infection
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Associate Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02000989
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Trauma Injury; Bone Infection
Keywords: ICG; Infection; Orthopedics; fluorescence imaging
MeSH Terms: conditions — Accidental Injuries; Infections | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic Infection: Subjects who have undergone previous orthopaedic trauma surgery and have developed and infection will be assessed for protocol inclusion criteria. Patients who meet all inclusion criteria and no exclusion criteria will be administered a single dose 2.5-5 mg/kg ICG dose intravenously ideally 24h prior to surgical debridement. Fluorescent images will be obtained pre and post irrigation and debridement
  Interventions: Procedure: imaging 24 hours following intravenous administration of ICG

INTERVENTIONS:
Procedure: imaging 24 hours following intravenous administration of ICG — Patients will be administered a single, FDA approved, ICG, 2.5-5mg/kg dose 24 hours prior to surgery. ICG fluorescence images will be acquired By a FDA approved surgical imaging device prior to surgical debridement. The wound will be irrigated as per standard procedure and another ICG fluorescence image will be acquired. The need for repeat debridement or tissue cultures will be left up to the treating surgeon.

SUMMARY:
The focus of this study is to (1) Explore variability in distribution of 24h ICG in bone and soft tissue infection (2) Evaluate the change in 24h ICG distribution from pre to post debridement (3) Preliminarily determine whether 24h ICG has the possibility predict infection / treatment failure. Patients will be administered a single, ICG, 2.5-5mg/kg dose 24 hours prior to surgery. The patient will be prepared and transported to surgery as per routine at Dartmouth-Hitchcock. ICG fluorescence images will be acquired prior to surgical debridement.

DETAILED DESCRIPTION:
Infection following trauma is one of the most prevalent and challenging complications faced by orthopedic surgeons in both military and civilian populations, occurring after up to 60% of open bone fractures. Several factors specific to this trauma place patients at high risk for infectious complications, including: traumatized tissues, open contaminated fracture, soft tissue coverage issues, catabolic state due to poly-trauma, prolonged hospitalization with exposure to nosocomial bacteria, and presence of metallic implants8. Infection requires one or more unplanned surgical procedures and leads to prolonged morbidity, loss of function, and potential loss of limb. Failed treatment for bone infection results in recurrent infection, requiring repeat surgical procedures in approximately 30% of patients.

Infection is known to display the enhanced permeability and retention effect with increased vascular permeability. Second window or 24h ICG represents an ideal method to identify these areas of increased vascular permeability. In some instances infected tissue can be hard to distinguish from healthy tissue when ICG is given immediately before optical imaging Second window ICG will allow surgeons to better distinguish infected tissue from healthy tissue as the ICG will have a better opportunity to permeate the infected tissue while it will have been expelled from the health tissue.

There are currently no accepted intraoperative tools that can be used to make objective decisions about which bone and tissue is infected and which is normal. Methods currently used to guide debridement are quite rudimentary. Clinical judgment is based on the gross appearance of soft tissue and bone, including color, turgor, and extent of soft tissue stripping. A burr may be used to look for bleeding bone. More extensive debridement is thought to minimize risk of index infection or reduce the rate of persistent infection; however, this comes at the cost of increasingly complex reconstructive procedures to fill bony defects. Clearly what is needed is a functional imaging system which can identify infected tissues to guide surgeons in the amount of tissue to debride. In turn, this will lead to fewer infections and a more effective treatment of SSIs at the fracture site. Both scenarios will allow patients to return to duty or work sooner.

The study endpoint is to determine the variability of bone and soft tissue perfusion in infection patients when given a single dose of ICG 24h prior to surgical debridement. The long term goal of this study is to aid in the development and optimization of bone specific imaging strategies that can be used to guide debridement and to optimize the quality of bone / tissue resection to minimize complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Extremity fracture.
3. Prior definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Superficial, deep, or organ space SSI (as per CDC criteria) at the fracture site that requires operative management.
5. Will have all planned SSI care surgeries performed by a participating surgeon or delegate.
6. Provision of informed consent.

Exclusion Criteria:

1. Fractures of the hand cannot be imaged.
2. Iodine allergy.
3. Burns at the SSI site.
4. Incarceration.
5. Expected survival of less than 90 days.
6. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
7. Adults unable to consent or whom do not have a LAR
8. Individuals who are not yet adults (infants, children, teenagers)
9. Pregnant or breastfeeding women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who have been diagnosed with an infection following orthopaedic trauma
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2024-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Orthopedic Infection
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Orthopedic Infection
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 71.5 [64 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Study Design Feasibility for Preoperative ICG Perfusion Rate as a Predictability Factor for Infection: Measured as Percentage of Patients With Analyzable Data
Description: This pilot study's objective is to preliminarily determine the study design feasibility of using a single dose of ICG given 24h preoperatively to predict recurrent infection/treatment failure. ICG Perfusion rates within the surgical site will be utilized to assess if there are any predictive measures that would indicate a higher risk of infection. Outcome measure is defined as the percentage of subjects with analyzable data.
Time Frame: Baseline
Measure: Number; unit: Percentage of subjects
Arm/Group | Orthopedic Infection
Number analyzed (Participants) | 2
Percentage of subjects | 0

ADVERSE EVENTS:
Time Frame: 6 months from study start
Description: per clinicaltrials.gov definitions
Arm/Group | Orthopedic Infection
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Due to low enrollment rates we were unable to provide significant results for the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT04927637/Prot_000.pdf
  • Informed Consent Form (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04927637/ICF_001.pdf